CLINICAL TRIAL: NCT06934499
Title: Clinical Observational Study on Tunisian Lung Cancer
Brief Title: Tunisian Lung Cancer Study
Acronym: LUNG-TUN
Status: Recruiting | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: The Multidisciplinary Consultation Meeting Thoracic Oncology of the Abderrahmen Mami Hospital (ROTHAM) (Unknown); Tunisian Society of Respiratory Diseases and Allergology (Unknown); Tunisian Society of Medical Oncology (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-01-LUNGTUN
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Cancer
Keywords: Pulmonary Cancer; Registry; Tunisia
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multicenter, observational, national study. Eligible patients will be recruited consecutively among subjects with proven lung cancer, including any disease stage withclinical, therapeutic and evolutive discription.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Patients receiving health care in the departments of pulmonology, oncology, radiation oncology and thoracic surgery, whose diagnosis is confirmed histologically and/or by cytology, at least 3 months before the inclusion date
* Informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants diagnosed with histologically confirmed lung cancer will be included in the study, regardless of sex, age, stage and histological subtype. Patients will be enrolled in the study consecutively The study will be conducted in different regions of Tunisia, encompassing several sites covering different departments in public hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1334 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic delay | Day 1
  Delay to set the pulmonary cancer diagnosis
Survival | 12 months
  Overall survival
Relapse | 12 months
  Time to relapse

SECONDARY OUTCOMES:
Recommendation Compliance | Day 1
  Compliance to national and international guidance of pulmonary cancer management

OTHER OUTCOMES:
Multidisciplinary Consultation Meetings | 12 months
  Number of Multidisciplinary Consultation Meetings

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Fenniche, MD, Study Chair — Multidisciplinary consultation meeting Thoracic of the Abderrahmen Mami ROTHA Hospital; Nesrine Mejri, MD, Study Chair — Multidisciplinary consultation meeting Thoracic of the Abderrahmen Mami ROTHA Hospital
Locations (2):
- Tunisia (2):
  - Tunisian Society of Medical Oncology, Aryanah
  - Tunisian Society of Respiratory Diseases and Allergology, Tunis

IPD SHARING:
Plan to Share IPD: No